CLINICAL TRIAL: NCT03764631
Title: Post-authorization Safety Study in Patients With Type 2 Diabetes Mellitus to Assess the Incidence of Ketoacidosis, Severe Complications of Urinary Tract Infection, Volume Depletion, and Dehydration Among Patients Treated With Empagliflozin or DPP-4 Inhibitors in Saudi Arabia
Brief Title: Post-authorization Safety Study in Type 2 Diabetic Patients in Saudi Arabia Treated With Empagliflozin to Assess the Incidence of Ketoacidosis, Severe Complications of Urinary Tract Infection, Volume Depletion, and Dehydration
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0149
Record Dates: First submitted 2018-11-26; First posted 2018-12-05 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Dipeptidyl Peptidase 4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subjects with Type 2 Diabetes mellitus
  Interventions: Drug: Empagliflozin; Drug: Dipeptidyl-peptidase 4 (DPP-4) inhibitors

INTERVENTIONS:
Drug: Empagliflozin — Drug
Drug: Dipeptidyl-peptidase 4 (DPP-4) inhibitors — Dipeptidyl-peptidase 4 - Drug

SUMMARY:
The objectives of this study are to assess the risk of ketoacidosis, severe urinary tract infections, volume depletion, and dehydration associated in patients with T2DM initiating Empagliflozin compared to patient initiating a dipeptidyl peptidase-4 (DPP-4) inhibitors over a 12-month period of follow-up, including the month of Ramadan

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed Informed consent form.
* The patients will be at least 18 years old at index date, diagnosed with Type 2 diabetes mellitus (T2DM) in Saudi Arabia, and who will initiate Empagliflozin or Dipeptidyl-peptidase 4 (DPP4) inhibitors treatment according to the local label and at the discretion of the treating physician during the study period, who have not used other sodium/glucose co-transporter 2 (SGLT2) or DPP4 inhibitors during the previous 12 months.

Exclusion Criteria:

* Known hypersensitivity to Empagliflozin, the comparator DPP-4 inhibitors or any of their excipients
* Patients for whom Empagliflozin or the comparator DPP-4 inhibitor is contraindicated according Saudi Food and Drug Authority (SFDA) approved label
* Patients prescribed fixed-dose combinations of SGLT2 inhibitors with DPP-4 inhibitors will be excluded.
* The same inclusion and exclusion criteria will be applied to the comparator group, which will include new users of DPP-4 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Main diagnosis for study entry
  -Patients diagnosed with T2DM will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1502 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mansour, +201028866717, Study Chair — ahmed.mansour@boehringer-ingelheim.com
Locations (21):
- Saudi Arabia (21):
  - Abha International Private Hospital, Abhā
  - DAFA Special Polyclinic, Jeddah
  - Ghassan Najeeb Pharaon Hospital, Jeddah
  - International Medical Center, Jeddah
  - Dr.Bakhsh Hospital, Jeddah
  - Dr. Soliman Fakeeh Hospital, Jeddah
  - Saudi German Hospital, Jeddah
  - Al Abeer Medical Center, Jeddah
  - Al-Abeer Medical Center, Jeddah
  - Al Abeer Polyclinic, Jeddah
  - Al Rahman Polyclinic, Mecca
  - Shifa Hospital, Mecca
  - Al-Noor Specialist Hospital, Mecca
  - Al Zafer Hospital, Najrān
  - Obesity, Endocrine and Metabolism Center, Riyadh
  - Riyadh Medical Center, Riyadh
  - Alalam Medical Center, Riyadh
  - Al Hada Armed Forces Hospital, Ta'if
  - Prince Fahad bin Sultan hospital, Tabuk
  - Al Amal Medical Group, Yanbu
  - Alansari Specialist Hospital, Yanbu

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. Studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement.

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A non-interventional study with new data collection from patients with type 2 diabetes mellitus in Saudi Arabia. The study used a "new users" design and compared new users of Empagliflozin to new users of Dipeptidyl peptidase-4 (DPP-4) inhibitors.
Pre-assignment Details: Only patients who met all of the inclusion and none of the exclusion criteria were enrolled into the study after signing the informed consent form.
Groups:
- Empagliflozin: Patients with type 2 diabetes mellitus (T2DM) and newly using Empagliflozin (e.g. Patients had not used other Sodium/Glucose co-transporter 2 (SLGT2) or Dipeptidyl peptidase-4 (DPP-4) inhibitors during the previous 12 months). Empagliflozin was administered according to the approved labels in Saudi Arabia. Patients were followed up for 12 months after the index date.
- DPP-4 Inhibitors: Patients with type 2 diabetes mellitus (T2DM) and newly using Dipeptidyl peptidase-4 (DPP-4) inhibitors (e.g. patients had not used other Sodium/Glucose co-transporter 2 (SLGT2) or DPP-4 inhibitors during the previous 12 months). DPP-4 inhibitors were administered according to the approved labels in Saudi Arabia. Patients were followed up for 12 months after the index date.
Period: Overall Study
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Started | 751 | 751
Completed | 710 | 698
Not Completed | 41 | 53
Not completed — Personal Reasons | 3 | 2
Not completed — Switching Therapy | 3 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 33 | 41
Not completed — No data as study site was closed | 2 | 6

BASELINE CHARACTERISTICS:
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in this study who signed the informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | DPP-4 Inhibitors | Total
Number analyzed (Participants) | 751 | 751 | 1502
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (10.3) | 52.9 (10.7) | 52.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273 | 264 | 537
  Male | 478 | 487 | 965
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ketoacidosis
Description: Ketoacidosis is defined as a serious complication of diabetes characterized by high levels of ketones in the body due to lack of insulin and low food intake.
Time Frame: Up to 12 months after the index date (defined as the date on which each identified new user received the index prescription for Empagliflozin or DPP-4 inhibitor).
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed the informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants | 1 | 1

2. Primary Outcome: Number of Participants With Severe Urinary Tract Infections (UTIs)
Description: Severe UTIs is defined as pyelonephritis or urosepsis.
Time Frame: Up to 12 months after index date (defined as the date on which each identified new user received the index prescription for Empagliflozin or DPP-4 inhibitor).
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed the informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Volume Depletion
Description: Volume depletion is defined as the reduction in the extracellular fluids.
Time Frame: as for outcome 2
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants | 6 | 7

4. Primary Outcome: Number of Participants With Dehydration
Description: Dehydration is defined as the loss of total body water that leads to hypertonicity.
Time Frame: as for outcome 2
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Ketoacidosis During Ramadan Periods
Description: Ketoacidosis is defined as a serious complication of diabetes characterized by high level of ketones in the body due to lack of insulin and low food intake.
  Ramadan period is defined as the first day of Ramadan to 29th day of Ramadan based on the Islamic Hijri calendar. The following Ramadan periods were included in this study:
  * Ramadan month 2019: 5. May to 4. Jun 2019 (± 1 to 2 days)
  * Ramadan month 2020: 23. April to 23. May 2020 (± 1 to 2 days).
Time Frame: Up to day 29.
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed the informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants
  Ramadan month 2019 | 0 | 0
  Ramadan month 2020 | 0 | 0

6. Secondary Outcome: Number of Participants With Severe Urinary Tract Infections (UTIs) During Ramadan Periods
Description: Severe UTIs is defined as pyelonephritis or urosepsis.
  Ramadan period is defined as the first day of Ramadan to 29th day of Ramadan based on the Islamic Hijri calendar. The following Ramadan periods were included in this study:
  * Ramadan month 2019: 5. May to 4. Jun 2019 (± 1 to 2 days)
  * Ramadan month 2020: 23. April to 23. May 2020 (± 1 to 2 days).
Time Frame: Up to day 29.
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed the informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants
  Ramadan month 2019 | 0 | 0
  Ramadan month 2020 | 0 | 0

7. Secondary Outcome: Number of Participants With Volume Depletion During Ramadan Periods
Description: Volume depletion is defined as the reduction in the extracellular fluids.
  Ramadan period is defined as the first day of Ramadan to 29th day of Ramadan based on the Islamic Hijri calendar. The following Ramadan periods were included in this study:
  * Ramadan month 2019: 5. May to 4. Jun 2019 (± 1 to 2 days)
  * Ramadan month 2020: 23. April to 23. May 2020 (± 1 to 2 days).
Time Frame: Up to day 29.
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed the informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants
  Ramadan month 2019 | 0 | 0
  Ramadan month 2020 | 0 | 0

8. Secondary Outcome: Number of Participants With Dehydration During Ramadan Periods
Description: Dehydration is defined as the loss of total body water that leads to hypertonicity.
  Ramadan period is defined as the first day of Ramadan to 29th day of Ramadan based on the Islamic Hijri calendar. The following Ramadan periods were included in this study:
  * Ramadan month 2019: 5. May to 4. Jun 2019 (± 1 to 2 days)
  * Ramadan month 2020: 23. April to 23. May 2020 (± 1 to 2 days).
Time Frame: Up to day 29.
Population: Enrolled Set: All patients with type 2 diabetes mellitus included in the study who signed the informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Number analyzed (Participants) | 751 | 751
Participants
  Ramadan month 2019 | 0 | 0
  Ramadan month 2020 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months.
Description: Enrolled Set: All patients with type 2 diabetes mellitus included in this study who signed the informed consent.
Arm/Group | Empagliflozin | DPP-4 Inhibitors
All-Cause Mortality (participants affected / at risk) | 0/751 | 0/751
Serious Adverse Events (participants affected / at risk) | 6/751 | 2/751
Other Adverse Events (participants affected / at risk) | 0/751 | 0/751
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin (N=751) | DPP-4 Inhibitors (N=751)
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT03764631/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT03764631/SAP_001.pdf